CLINICAL TRIAL: NCT07357779
Title: Clinical Efficacy and Health Economic Evaluation of an Intelligent Diagnostic and Treatment Model Based on Digital Cognitive Behavioral Therapy for Insomnia Disorder
Brief Title: Clinical Efficacy and Health Economic Evaluation of an Intelligent Diagnostic and Treatment Model
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zan Wang (Other)
Responsible Party: Sponsor-Investigator, Zan Wang, Sleep Center Director, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBTI-V1
Record Dates: First submitted 2026-01-04; First posted 2026-01-22 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional treatment group (Sham Comparator)
  Interventions: Drug: Traditional treatment
- Intelligent diagnosis and treatment group (Active Comparator)
  Interventions: Other: Intelligent Diagnostic and Treatment Model

INTERVENTIONS:
Other: Intelligent Diagnostic and Treatment Model — Intelligent CBTI
  Arms: Intelligent diagnosis and treatment group
Drug: Traditional treatment — sleep drug treatment
  Arms: Traditional treatment group

SUMMARY:
The purpose of this study is to evaluate the clinical and cost-effectiveness of an intelligent therapy based on digital cognitive behavioral therapy for insomnia disorders

DETAILED DESCRIPTION:
Insomnia is a highly prevalent and distressing disorder, yet access to its first-line treatment, cognitive behavioral therapy for insomnia (CBT-I) remains highly limited. Therefore, providing accessible and personalized CBT-I is pivotal in its application. With the widespread development of the internet and mobile application devices, digital Cognitive Behavioral Therapy for Insomnia (dCBT-I) has opened new avenues for the diagnosis and treatment of insomnia disorder. Studies have explored internet-based, self-administered CBT-I treatment models, which have increased access to effective psychological therapy for patients with insomnia.

ELIGIBILITY:
Inclusion Criteria:

* (1) Clinical diagnosis of insomnia disorder; (2) Cooperate to complete the questionnaire surveys.

Exclusion Criteria:

* (1) Current use of central nervous system stimulants; (2) Use of analgesics, theophylline preparations, steroid medications; (3) Alcohol abuse or regular alcohol intake; (4) Diagnosis of other sleep disorders (e.g., obstructive sleep apnea, rapid eye movement sleep behavior disorder, restless legs syndrome) ; (5) Sleep disorders secondary to organic diseases (e.g., epilepsy, diabetes, renal failure).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
the score of Insomnia Severity Index scale | 6 weeks and 3 months
  The total score ranges from 0 to 28, and a higher score indicates higher levels of insomnia severity. A score of 8 or greater is the cut point for clinically possible insomnia
the score of 7-item Generalized Anxiety Disorder scale | 6 weeks and 3 months
  The total score ranges from 0 to 21, and a higher score indicates higher levels of anxiety symptoms. A score of 10 or greater is the cut point for clinically possible anxiety
the score of Patient Health Questionnaire-9 scale | 6 weeks and 3 months
  The total score ranges from 0 to 27, and a higher score indicates higher levels of depression symptoms. A score of 10 or greater is the cut point for clinically possible depression symptom
the value of European Quality of Life Five Dimension | 6 weeks and 3 months
  The European Quality of Life Five Dimension is a standardized measure of health-related quality of life assessing five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Higher scores indicate better quality of life
the value of Work Productivity and Activity Impairment: General Health | 6 weeks and 3 months
  The Work Productivity and Activity Impairment: General Health (WPAI:GH) questionnaire assesses the impact of health problems on work productivity and daily activities over the past seven days, including absenteeism, presenteeism, overall work productivity loss, and activity impairment. Scores are expressed as percentages, with higher scores indicating greater impairment
the value of direct medical costs | 6 weeks and 3 months
  Direct medical costs refer to healthcare expenditures incurred by patients during visits to medical institutions, including consultation fees, diagnostic and examination costs, medication expenses, and hospitalization costs

SECONDARY OUTCOMES:
Change in plasma corticotropin-releasing factor (CRF) level | 6 weeks and 3 months
  Plasma corticotropin-releasing factor (CRF) concentration was measured as a biomarker of hypothalamic-pituitary-adrenal (HPA) axis activity. Higher levels indicate increased neuroendocrine stress response. Unit of Measure: pg/mL
Change in plasma cortisol level | 6 weeks and 3 months
  Plasma cortisol concentration was assessed as an indicator of hypothalamic-pituitary-adrenal (HPA) axis function. Higher levels reflect increased physiological stress response. Unit of Measure: μg/dL
Change in serum interleukin-6 (IL-6) level | 6 weeks and 3 months
  Serum interleukin-6 (IL-6) concentration was measured as a marker of systemic inflammation. Higher levels indicate greater inflammatory activity. Unit of Measure: pg/mL
Change in serum brain-derived neurotrophic factor (BDNF) level | 6 weeks and 3 months
  Serum brain-derived neurotrophic factor (BDNF) concentration was measured as a biomarker associated with neuroplasticity and neuronal function. Higher levels indicate enhanced neurotrophic activity. Unit of Measure: pg/mL
Change in total sleep time (TST) measured by polysomnography | 6 weeks and 3 months
Change in sleep onset latency (SOL) measured by polysomnography | 6 weeks and 3 months
Change in wake after sleep onset (WASO) measured by polysomnography | 6 weeks and 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided